CLINICAL TRIAL: NCT07087236
Title: Sedentary Activities and Passive-to-Intense Effects on Neuro-Cognitive States
Acronym: SAPIENS
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Valparaiso (Other)
Responsible Party: Principal Investigator, Carlos Cristi Montero, Principal Investigator, Pontificia Universidad Catolica de Valparaiso
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BIOEPUCV-H 858-2024
Record Dates: First submitted 2025-07-06; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Cognition; Sedentary Behaviors
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: This intra-individual study will be conducted in three separate days. The first day will be performed the "familiarization day" for those being evaluated, assessing basal (through spontaneous sitting activity) and maximal (through N-back test) cognitive load and additionally, the evaluators will conducted physical measures (e.g., body composition through DEXA, fitness by the 3-minute step and strength using dynamometer (Jamar Plus + Digital Hand Dynamometer, Sammons Preston, USA), and sociodemographic questionnaire. The second day, the evaluators will conduct four randomized activities. Finally, the third day, the evaluators will conduct the final 3 activities, which also will be randomized between mentally passive and active activities.
Who Masked: Participant, Investigator
Masking Description: Doble-blind. Both participants and the statistician were blinded to the intervention condition; however, the assessors administering the activities were not blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Baseline Cognitive Condition (Active Comparator)
  Interventions: Behavioral: Baseline Cognitive Load
- Maximum Cognitive Load Condition (Active Comparator)
  Interventions: Behavioral: Maximum Cognitive Load
- Experimental Mentally Active and Mentally Passive Sedentary Activities (Experimental)
  Interventions: Behavioral: Mental active/pasive activities

INTERVENTIONS:
Behavioral: Maximum Cognitive Load — Participants will perform a working memory task (through N-back 1-to-3) to evaluate the upper limit of cognitive demand.
  Arms: Maximum Cognitive Load Condition
Behavioral: Mental active/pasive activities — Participants will engage in 7 activities, presented in a randomly assigned order across two separate days, to assess their impact on cognitive load:
  1. playing a videogame (Tetris ®)
  2. listening a podcast (including a final question)
  3. watching a documentary (including a final question)
  4. reading a document extract (including a final question)
  5. watch a reality show extract (including a final question)
  6. listening music, they like it
  7. scrolling their Tik-Tok/Instagram
  Arms: Experimental Mentally Active and Mentally Passive Sedentary Activities
Behavioral: Baseline Cognitive Load — Participants will sit quietly for 5 minutes to establish baseline spontaneous neurophysiological parameters.
  Arms: Baseline Cognitive Condition

SUMMARY:
Prolonged sedentary behavior is linked to poorer metabolic health, yet its effect on cognitive load and brain function remains unclear. Evidence indicates that "mentally active" sedentary tasks (e.g., reading) may support cognition, whereas "mentally passive" tasks (e.g., scrolling social media) may impair it. The cognitive demands associated with these behaviors across the general population are still poorly defined. This project will compare the acute neurophysiological and perceptual responses elicited by mentally active versus passive sedentary tasks across various age groups and in individuals with specific health conditions (i.e., obesity), clarifying how these behaviors differ in the cognitive load they impose. Neuro-cognitive, physiological, and perceptual responses will be assessed with a multimodal battery that includes portable electroencephalography combined with functional near-infrared spectroscopy (EEG + fNIRS; MUSE), eye-tracking (Pupil Core), alertness and visual fatigue via critical flicker fusion testing (CFFT; Lafayette Instrument), autonomic balance through heart-rate variability (HRV) recorded with a Polar H10 monitor, and the self-reported cognitive load assessed using the NASA Task Load Index (NASA-TLX). We hypothesise that mentally passive sedentary activities will elicit a lower cognitive load than mentally active tasks. By comparing different age groups and health conditions within a single protocol, the study will generate an initial set of group-specific data; subsequent independent studies can build on these findings to explore moderation effects in greater depth. Collectively, the results will provide both the theoretical rationale and the empirical evidence needed to sustain the "mentally active" versus "mentally passive" terminology in sedentary-behaviour research, with the ultimate aim of improving mental and cognitive health.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 5 to 17 years, attending school.
* Adults aged 18 and above, without an upper age limit.
* Participants with and without specific health conditions, such as obesity.
* Ability to perform sedentary activities and comprehend instructions.

Exclusion Criteria:

* Severe visual impairments affecting reading or text visualization.
* Use of conventional glasses and history of migraine or epilepsy (due to preventive request for the flicker fusion test)
* Current use of medications that significantly influence cognitive function (unless the health condition being evaluated requires it).
* Other conditions interfering with cognitive or neurophysiological assessments.

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Electroencephalography-derived cortical activity (EEG) | Day 1 and 2
  This outcome will be evaluated using a portable EEG system (MUSE Athena), which will evaluate four types of brain waves-alpha (8-12 Hz), gamma (31-90 Hz), theta (4-7 Hz), and beta (13-30 Hz)-along with two wave ratios: theta/alpha and beta/alpha.
Hemodynamic Response (fNIRS) | Day 1 and 2
  This outcome will be evaluated using a portable functional near-infrared spectroscopy system (fNIRS) in the MUSE headband, assessing changes in oxyhemoglobin (HbO) and deoxyhemoglobin (HbR) concentrations in the prefrontal cortex.
Eye-Tracking Metrics | Day 1 and 2
  This outcome will be evaluated using a validated portable eye tracker (Pupil Core) to assess eye metrics.
Heart Rate Variability (HRV) | Day 1 and 2
  This outcome will be evaluated using a chest strap device connected wirelessly to a tablet (Polar H10). Changes in HRV and heart rate are analyzed as a physiological marker (autonomic balance).
Critical Flicker Fusion Threshold (Flicker Fusion) | Day 1 and 2
  This outcome will be evaluated using the Flicker Fusion System (Lafayette Instrument Company) with the "coincident" stimulus to determine the critical flicker fusion threshold (Hz).
Self-Reported Cognitive Load (NASA-TLX) | day 2
  The Self-Reported Cognitive Load is measured using the NASA Task Load Index (NASA-TLX). Scores range from 0 to 100, with higher scores indicating greater cognitive load. Capturing subjective workload across six dimensions: mental demand, physical demand, temporal demand, effort, performance, and frustration.

CONTACTS AND LOCATIONS:
Locations (1):
- Pontificia Universidad Católica de Valparaíso, Viña del Mar, Chile